CLINICAL TRIAL: NCT04459299
Title: An Evaluation of Performance of the CorPath® GRX System in Robotic-PCI During Acute STEMI
Brief Title: CorPath GRX STEMI Study
Acronym: TREAT GRX
Status: Terminated | Type: Observational
Why Stopped: Low enrollment and sponsor business decision
Sponsor: Corindus Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 104-09062
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2022-01

CONDITIONS: STEMI - ST Elevation Myocardial Infarction; CAD
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- STEMI patients with clinical indication for primary PCI: Subjects with a clinical indication of STEMI.
  Interventions: Device: Robotic-PCI (CorPath GRX System)

INTERVENTIONS:
Device: Robotic-PCI (CorPath GRX System) — Robotic-PCI for acute ST elevation myocardial infarction (STEMI).

SUMMARY:
This study will evaluate the performance of the CorPath GRX System in Robotic Primary PCI (RPPCI) in the treatment of ST-elevated myocardial infarction (STEMI).

DETAILED DESCRIPTION:
This is a prospective, post-market, single-arm, multi-center, observational study to evaluate the performance of the CorPath GRX System during robotic-PCI for acute ST elevation myocardial infarction (STEMI).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤ 80 years
* Patients with STEMI<12 h of symptom onset
* Patient deemed appropriate for robotic-assisted PCI
* The subject has been informed of the nature of the study, agrees to its provisions, and has provided written consent

Exclusion Criteria:

Cardiogenic shock

* Cardiac arrest
* Need for manual or mechanical thrombectomy
* Failure/inability/unwillingness to provide informed consent
* The Investigator determines that the subject or the coronary anatomy is not suitable for robotic-assisted primary PCI treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a clinical indication of STEMI.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2020-11-26 (Actual); Study Completion 2020-11-29 (Actual)

PRIMARY OUTCOMES:
Time from Catheterization Lab Arrival to Device Activation (CLADA) by CorPath GRX System. | Procedure
  Time measured from arrival to Cath Lab to device activation by CorPath GRX System.

SECONDARY OUTCOMES:
Freedom from MACE events | 72-hours
  Completion of the STEMI procedure without in-hospital major adverse cardiovascular event MACE). MACE is defined as cardiac death, clinically driven target vessel revascularization (TVR) by repeat PCI, surgical bypass for any segment of the target vessel or stent thrombosis.
First Medical Contact (FMC) to device activation time | Procedure
  Time at which first patient evaluation.
Access to device activation | Procedure
  Time measured from access sheath insertion to device activation by CorPath GRX System.
Access to wire time | Procedure
  Defined as time measured from sheath insertion to crossing the lesion with the coronary guidewire.
Overall procedure time | Procedure
  Defined as the time measured from sheath insertion to removal of the last device used to treat the culprit lesion.
Fluoroscopy time | Procedure
  Total fluoroscopy time (min.) utilized during the procedure as recorded by the Imaging System.
Patient radiation exposure | Procedure
  DAP (dose-area-product) and AK (air kerma) as recorded during the procedure.
Contrast fluid volume | Procedure
  Total contrast volume (mL/cc) used during the procedure.
Conversion to manual (Binary) | Procedure
  Conversion from robotic technique to manual technique due to inability to successfully wire lesion or deliver first device.
Technical success | Procedure
  Completion of the PCI procedure entirely robotically or with partial manual assistance.
Serious adverse events | 72-hours
  All Serious Adverse Events (SAEs) from the start of the CorPath GRX procedure until the end of the study will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore F Mannino, DO, MA, Study Chair — WellStar Health System
Locations (1):
- Wellstar Kennestone Hospital, Marietta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available 12 months after study completion.

REFERENCES:
- [Background] Hirshfeld JW Jr, Balter S, Brinker JA, Kern MJ, Klein LW, Lindsay BD, Tommaso CL, Tracy CM, Wagner LK, Creager MA, Elnicki M, Lorell BH, Rodgers GP, Weitz HH; American College of Cardiology Foundation; American Heart Association/; HRS; SCAI; American College of Physicians Task Force on Clinical Competence and Training. ACCF/AHA/HRS/SCAI clinical competence statement on physician knowledge to optimize patient safety and image quality in fluoroscopically guided invasive cardiovascular procedures: a report of the American College of Cardiology Foundation/American Heart Association/American College of Physicians Task Force on Clinical Competence and Training. Circulation. 2005 Feb 1;111(4):511-32. doi: 10.1161/01.CIR.0000157946.29224.5D. No abstract available. PMID 15687141
- [Background] Klein LW, Miller DL, Balter S, Laskey W, Haines D, Norbash A, Mauro MA, Goldstein JA; Joint Inter-Society Task Force on Occupational Hazards in the Interventional Laboratory. Occupational health hazards in the interventional laboratory: time for a safer environment. Catheter Cardiovasc Interv. 2009 Feb 15;73(3):432-8. doi: 10.1002/ccd.21801. PMID 19214981
- [Background] Miller DL, Schueler BA, Balter S; National Council on Radiation Protection and Measurements; International Commission on Radiological Protection. New recommendations for occupational radiation protection. J Am Coll Radiol. 2012 May;9(5):366-8. doi: 10.1016/j.jacr.2012.02.006. No abstract available. PMID 22554637
- [Background] Ciraj-Bjelac O, Rehani MM, Sim KH, Liew HB, Vano E, Kleiman NJ. Risk for radiation-induced cataract for staff in interventional cardiology: is there reason for concern? Catheter Cardiovasc Interv. 2010 Nov 15;76(6):826-34. doi: 10.1002/ccd.22670. PMID 20549683
- [Background] Vano E, Kleiman NJ, Duran A, Romano-Miller M, Rehani MM. Radiation-associated lens opacities in catheterization personnel: results of a survey and direct assessments. J Vasc Interv Radiol. 2013 Feb;24(2):197-204. doi: 10.1016/j.jvir.2012.10.016. Epub 2013 Jan 28. PMID 23369556
- [Background] Mahmud E, Naghi J, Ang L, Harrison J, Behnamfar O, Pourdjabbar A, Reeves R, Patel M. Demonstration of the Safety and Feasibility of Robotically Assisted Percutaneous Coronary Intervention in Complex Coronary Lesions: Results of the CORA-PCI Study (Complex Robotically Assisted Percutaneous Coronary Intervention). JACC Cardiovasc Interv. 2017 Jul 10;10(13):1320-1327. doi: 10.1016/j.jcin.2017.03.050. PMID 28683937

DOCUMENTS (1):
  • Study Protocol (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/99/NCT04459299/Prot_000.pdf